CLINICAL TRIAL: NCT06585631
Title: The Collaborative Care PrTNER (Prevention, Treatment, Navigation, Engagement, Resource) Project
Brief Title: The Collaborative Care PrTNER Study
Acronym: PrTNER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Johns Hopkins University (Other); Baltimore City Health Department (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 23-021859; R01DA059022 (NIH)
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: HIV; Substance Use Disorders; Substance Use; AIDS
Keywords: Gay, Bisexual; Young men who have sex with men; Young Black men who have sex with men; Young Latino men who have sex with men; HIV; AIDS; Substance use; Substances use disorder; men who have sex with men; young gay men; gay men; drug use; alcohol use; preexposure prophylaxis; PrEP; peer coaches; community health worker; LGBT; bisexual
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Homosexuality; Bisexuality; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: YBLMSM will be randomized (1:1) to intervention vs. SOC for each aim, using a computer-stratified randomization to yield balanced randomization between younger (15-19) and older (20-24) age groups and based on substance use risk as determined by their screener questionnaire. A separate stratum will be defined for each combination of covariates (age group and substance use risk) and participants will be randomized to Participants will sign a release of medical information for HIV/SU/Mental Health Disorders outcomes. Visits occur at baseline (time 0), 3, 6, 9, and 12 months. Participants will complete an interviewer-administered, electronic baseline and quarterly surveys followed by the collection of samples for biologic measures. Survey assess individual, interpersonal, multi-level barriers to HIV prevention care and treatment in the community, and structural levels. The survey will identify varying severity of hazardous/harmful substance use and co-existing mental health needs.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants randomized to CC PrTNER will be assigned a peer coach, complete interviewer-administered behavioral surveys, receive psychoeducation, identify health goals.
  Interventions: Behavioral: CC PrTNER
- Standard of Care (No Intervention): The participant's provider will receive an electronic alert in real time of the participant's positive screen for SU and a list of area substance treatment resources. The provider at their discretion will provide counseling or initiate a referral to in-clinic or community-based resources for SU assessment and treatment. Each of our clinical sites has case management resources for counseling and support for linkage to co-located SU treatment or community-based resources for inpatient or outpatient SU treatment as indicated at the discretion of the HIV/PrEP provider. SOC arm participants will not be assigned a coach. Study visit surveys and sample collection at baseline, 3, 6, 9, and 12 months are identical for intervention and SOC arm participants. Research personnel will make no attempts to provide brief intervention, motivational interviewing (MI), or case management.

INTERVENTIONS:
Behavioral: CC PrTNER — Participants randomized to CC PrTNER will be assigned a peer coach. They will conduct interviewer-administered behavioral surveys. The surveys provide an in-depth assessment of SU, HIV prevention and care, engagement, and adherence. Behavioral surveys are administered monthly. The coach will discuss with the participant the areas that are flagged by the psychiatrist; provide psychoeducation around areas identified, and work with the participant to identify their health goals and how changes in SU may help feed into self-defined goals. The coach will meet weekly with the consultant addiction psychiatrist who will make a provisional diagnosis and define a treatment plan with clear goals for treatment outcome. Recommendations will be communicated electronically to the HIV or PrEP provider to facilitate implementation. The coach utilizes MI skills to implement the individually tailored to facilitate the adoption and maintenance of health behaviors.
  Arms: Intervention

SUMMARY:
A randomized controlled trial to assess the ability of a Collaborative Care Prevention, Treatment, Navigation, Engagement, Resource (PrTNER) intervention to increase initiation of preexposure prophylaxis (PrEP) (for those at-risk for HIV) and decrease viral load (for those living with HIV) among young Black and Latino men who have sex with men (YBLMSM) aged 15 to 24 through engagement in SU treatment.

DETAILED DESCRIPTION:
The Collaborative Care (CC) PrTNER is a multi-component intervention developed by members of the research team specifically for YBLMSM aged 15 to 24 who are at-risk for or living with HIV. This model moves beyond the individual to consider the broader context in which, substance use (SU), and HIV risk are (re)produced.

Enhanced models that integrate SU treatment into HIV and PrEP primary care services (using a collaborative care approach that incorporates feedback from a psychiatrist and support from a peer coach) are needed to address the nuance of substance use in this population. We, therefore, are proposing to conduct a randomized trial to evaluate an integrated collaborative care model (CC PrTNER).

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

* 15-24 years old;
* Cisgender male;
* Self-identified Black/African American race or Latino/Hispanic ethnicity;
* Report prior oral/anal sex with another male;
* At-risk for HIV (condomless anal sex or positive sexually transmitted infection (STI) in last 6 months);
* Moderate-to-high risk SU behaviors based upon a Car, Relax, Alone, Forget, Friends, Trouble (CRAFFT) score ≥2,
* Living in Philadelphia, PA or Baltimore, MD, and surrounding areas;
* Able to read and write in English

Aim 2:

* 15-24 years old;
* Cisgender male;
* Self-identified Black/African American race or Latino/Hispanic ethnicity;
* Report prior oral/anal sex with another male;
* Living with a diagnosis of HIV;
* CRAFFT score ≥2,
* Living in Philadelphia, PA or Baltimore, MD, and surrounding areas;
* Able to read and write in English

Aim 3

• All randomized study participants will be included in Aim 3.

Exclusion Criteria:

Aim 2:

* Participants will be excluded if they are:
* Assigned female sex at birth
* Identify as transgender
* Outside the age criteria (<15 or >24 years old)
* Cognitively unable to complete study requirements
* Living outside of the two geographic areas
* Do not screen positive for SU
* No prior substance use history
* No prior oral or anal sex;
* Unable to read or write in English,
* Plan to move in the next 12 months.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — cis-gender young men
Enrollment: 275 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
PrEP uptake at 12 months | 12 months
  PrEP uptake from baseline to 12 month survey. Biomedical assessment of PrEP use at 12 months, Intraerythrocytic Tenofovir-Diphosphate (TVF-DP) from dried blood spot (DBS) >700 fmol/punch (oral PrEP), 2+ on-time injections of Long-acting injectable cabotegravir (CAB-LA)
HIV virologic suppression at 12 months | 12 months
  Viral load < 20 copies/mL from baseline to 12 months
Number of days of past-28-day non-tobacco drug/alcohol use | 12 months
  Number of days of past-28-day non-tobacco drug/alcohol use, assessed via Timeline Followback Method Assessment (TLFB) from baseline to 12 months

SECONDARY OUTCOMES:
PrEP persistence | 12 months
  Duration of time participants maintain benchmark TFV-DP concentrations from baseline to 12 months
Sustained viral suppression | 12 months
  Duration of time participants are virally suppressed from baseline to 12 months
Uptake of HIV Antiretroviral therapy (ART) treatment | 12 months
  Frequency of inadequate drug measurements and drug-resistant virus in those who are not virally suppressed from baseline to 12 months
Mean number of negative urine drug screens (UDS) | 12 months
  Mean number of negative UDS at 12 months
Substance-related problems | 12 months
  Substance-related problems as defined by Alcohol Use Disorders Identification Test (AUDIT), Cannabis Use Disorders Identification Test - Revised (CUDIT-R), and Severity of Dependence Scale (SDS scores) from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Renata Sanders, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Johns Hopkins Center for Adolescent and Young Adult Health, Baltimore, Maryland
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared between sites and made available to other NIH funded researchers upon approval of written official request and shared via applicable Johns Hopkins University Data Transfer Agreements. No data will be released that would allow the identification of any respondent, unless written informed permission for this is obtained.
  Data will also be shared with key stakeholders throughout the study, between sites, and made available to study participants after the analysis is completed. We will summarize and present findings in a summary report, webinar, and in a face-to-face meeting at each site once analyses are completed. The summary report will be emailed to participants, including, adolescents, providers, and community partners about the findings of the work. As part of the Center for AIDS Research (CFAR) Initiatives, we will share our findings and data, when appropriate, with the Baltimore and Philadelphia CFARs and Ryan White sites.
Time Frame: Data will be shared between sites and with key stakeholders throughout the study. At the conclusion of the study data will be made available to participants.
Access Criteria: Applicable Johns Hopkins University Data Transfer Agreements